CLINICAL TRIAL: NCT06707779
Title: Effect of Proprioceptive Neuromuscular Facilitation With and Without Electrical Stimulation on Pain and Functional Disability in Patients With Chronic Lumbar Radiculopathy
Brief Title: PNF With and Without Electrical Stimulation in Patients With Chronic Lumbar Radiculopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/24/0214 Azka Yaseen
Record Dates: First submitted 2024-11-25; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Lumbar Radiculopathy
Keywords: pain; disability
MeSH Terms: conditions — Radiculopathy; Pain | interventions — Electric Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PNF with electrical stimulation (Experimental): participants in this arm receive PNF with electrical stimulation to reduce pain and functional disability in patients with chronic lumbar radiculopathy
  Interventions: Other: PNF with electrical stimulation
- PNF without electrical stimulation (Experimental): participants in this arm receive PNF without electrical stimulation to reduce pain and functional disability in patients with chronic lumbar radiculopathy
  Interventions: Other: PNF without electrical stimulation

INTERVENTIONS:
Other: PNF with electrical stimulation — Group A receive PNF including combination of isotonic and rhythmic stabilization on trunk with electrical stimulation Participants perform three sets10 repetitions at maximal resistance The resting interval of 30 seconds and 60 seconds will be provided after the completion of 10 repetitions for each pattern and between sets respectively.
  In total all PNF exercise will be held for 30 to 45 minutes. 'BURST' TENS (acupuncture-like TENS), characterized by discontinuous stimulation at low frequencies (1-4 Hz), with wave durations of 100-400 ms and high intensities, inducing weak muscle twitches for 10 minutes.
  Arms: PNF with electrical stimulation
Other: PNF without electrical stimulation — Group B receive PNF including combination of isotonic and rhythmic stabilization on trunk without electrical stimulation. Participants perform three sets of 10 repetitions at maximal resistance will be provided by the same physiotherapist.
  The resting interval of 30 seconds and 60 seconds will be provided after the completion of 10 repetitions for each pattern and between sets respectively.
  In total all PNF exercise will be held for 30 to 45 minutes.
  Arms: PNF without electrical stimulation

SUMMARY:
Numerous researches have shown how PNF is been used to treat non specific low back pain, subacromial impingement, cervical radiculopathy and many others. In some studies different techniques like Mckenzie method, spinal mobilization and Mulligan traction other than PNF were being used to treat lumbar radiculopathy. According to researchers knowledge little literature available to see the effectiveness of PNF with electrical stimulation in patients with chronic lumbar radiculopathy. Therefore, the purpose of the current study is to examine the effects of PNF with electrical stimulation in patients with chronic lumbar radiculopathy.

ELIGIBILITY:
Inclusion Criteria:

* • Diagnosed cases of lumbar radiculopathy

  * Either one or both legs affected by radiating pain
  * Signs of nerve root compression like paresthesia, numbness, tingling, sharp pain
  * Impaired deep tendon reflex(knee jerk, ankle jerk)
  * Both male and female
  * Radiological evidence of lumbar spondylosis with radiculopathy
  * Age group between 40 to 70 years
  * Positive SLR test between 45° to 70°
  * All subjects with symptoms for duration of more than 6 weeks
  * Increase leg pain by coughing and sneezing

Exclusion Criteria:

* Serious spinal conditions e.g infection, tumor, osteoporosis
* Uncontrolled hypertension
* Severe cognitive impairment
* Other neurological conditions and systemic illness like kidney and visceral diseases
* Vertebral fracture and spondylolisthesis
* Pregnant women
* History of spinal surgery in previous 6 months
* Clinical conditions such as oversensitive skin, patients with cardiac pacemakers where application of TENS is contraindicated

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2024-02-02 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
pain numeric rating scale | 6th week
  The pain numeric rating scale is a segmented numeric version of visual analog scale in which a respondent selects a whole number 0 to 10 that reflects the intensity of pain. The 11 point numeric scale ranges from 0 representing no pain and 10 representing extreme pain. Higher scores indicating greater pain intensity. e.g. as bad as you can imagine or worst pain. NPRS takes less than 1 minute to complete and easy to administer and score.
Modified Oswestry disability index | 6th week
  MODI also known as the Oswestry Low Back Pain Disability Questionnaire, as a very crucial instrument to assess a patient's functional disability over the long term. MODI is a patient completed questionnaire included 10 sections of questions. This tool is effective for persistent severe disability. The MODI domains are the following: pain intensity, personal care, lifting, walking, sitting, standing, sleeping, social life, travelling and employment/home making. Each section has six statements that are scored from 0 means minimum degree of difficulties in that activity to 5 means maximum degree of difficulty.

CONTACTS AND LOCATIONS:
Overall Officials: Arnab Altaf, PP DPT, Principal Investigator — Riphah International University Lahore
Locations (1):
- Amin welfare and teaching hospital , Awan center, Sialkot, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaya DO, Celenay ST, Secer E, Biceroglu H. Pain intensity, spine structure, and body composition in patients with acute discogenic lumbar radiculopathy. Musculoskelet Sci Pract. 2024 Oct;73:103133. doi: 10.1016/j.msksp.2024.103133. Epub 2024 Jul 2. PMID 38968681
- [Background] Moustafa IM, Diab AAM, Harrison DE. Does Improvement towards a Normal Cervical Sagittal Configuration Aid in the Management of Lumbosacral Radiculopathy: A Randomized Controlled Trial. J Clin Med. 2022 Sep 29;11(19):5768. doi: 10.3390/jcm11195768. PMID 36233636
- [Background] Clark R, Weber RP, Kahwati L. Surgical Management of Lumbar Radiculopathy: a Systematic Review. J Gen Intern Med. 2020 Mar;35(3):855-864. doi: 10.1007/s11606-019-05476-8. Epub 2019 Nov 11. PMID 31713029
- [Background] Ghasabmahaleh SH, Rezasoltani Z, Dadarkhah A, Hamidipanah S, Mofrad RK, Najafi S. Spinal Manipulation for Subacute and Chronic Lumbar Radiculopathy: A Randomized Controlled Trial. Am J Med. 2021 Jan;134(1):135-141. doi: 10.1016/j.amjmed.2020.08.005. Epub 2020 Sep 13. PMID 32931763
- [Background] Samant P, Tawde P, Tawde DN. Understanding How Patients With Lumbar Radiculopathy Make Sense of and Cope With Their Symptoms. Cureus. 2024 Mar 26;16(3):e56987. doi: 10.7759/cureus.56987. eCollection 2024 Mar. PMID 38665744
- [Background] Pojskic M, Bisson E, Oertel J, Takami T, Zygourakis C, Costa F. Lumbar disc herniation: Epidemiology, clinical and radiologic diagnosis WFNS spine committee recommendations. World Neurosurg X. 2024 Feb 20;22:100279. doi: 10.1016/j.wnsx.2024.100279. eCollection 2024 Apr. PMID 38440379